CLINICAL TRIAL: NCT06554184
Title: A Randomized Phase III Study Evaluating the Efficacy and Safety of HR20013 for Nausea and Vomiting Associated With Moderate Emetic Risk Anticancer Agents
Brief Title: HR20013 for Nausea and Vomiting Associated With Moderate Emetic Risk Anticancer Agents
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fujian Shengdi Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HR20013-302
Record Dates: First submitted 2024-08-13; First posted 2024-08-15 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-10

CONDITIONS: Nausea and Vomiting Associated With Moderate Emetic Risk Anticancer Agents
MeSH Terms: conditions — Nausea | interventions — Dexamethasone; Palonosetron

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HR20013 + dexamethasone + palonosetron placebo (Experimental)
  Interventions: Drug: HR20013 + dexamethasone + palonosetron placebo
- Palonosetron + dexamethasone + HR20013 placebo (Active Comparator)
  Interventions: Drug: Palonosetron + dexamethasone + HR20013 placebo

INTERVENTIONS:
Drug: HR20013 + dexamethasone + palonosetron placebo — HR20013 + dexamethasone + palonosetron placebo
  Arms: HR20013 + dexamethasone + palonosetron placebo
Drug: Palonosetron + dexamethasone + HR20013 placebo — Palonosetron + dexamethasone + HR20013 placebo
  Arms: Palonosetron + dexamethasone + HR20013 placebo

SUMMARY:
This study is aimed to evaluate the efficacy and safety of HR20013 versus palonosetron for nausea and vomiting associated with moderate emetic risk anticancer agents

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older, of either gender
2. Has a histologically or cytologically confirmed malignant disease
3. Naïve to cytotoxic chemotherapy
4. Scheduled to receive first course of moderate emetic risk anticancer agents
5. Predicted life expectancy of ≥ 3 months
6. Has a performance status (ECOG scale) of 0 to 1
7. Adequate organ function
8. female subjects of childbearing potential must have a negative blood pregnancy test within 72 hours before randomization; and must be non-lactating;
9. Able and willing to provide a written informed consent

Exclusion Criteria:

1. Received or planned to receive total body irradiation, or radiation therapy to the abdomen, pelvis, Whole brain and spinal cord, head and neck , or chest within 7 days before randomization or within Days 1 to 8 of treatment
2. Scheduled to receive any moderate emetic risk anticancer agents from Day 1 to 6
3. Planned to receive treatment with a chemotherapy regimen including ordinary paclitaxel (with castor oil as solvent);
4. Medications with potential antiemetic efficacy within 2 days before randomization;
5. Began using opioids within 7 days prior to randomization or had a dose adjustment within the last 7 days.
6. Systemic corticosteroid therapy or sedative antihistamines within 7 days before randomization;
7. Use of palonosetron within 14 days before randomization;
8. Use of NK-1 receptor antagonists within 28 days before randomization;
9. Use of moderate to strong CYP3A4 inhibitors within 7 days before randomization; use of moderate to strong CYP3A4 inducers or specific CYP2D6 substrates within 28 days before randomization;
10. Vomiting and/or retching and nausea within 24 hours before randomization;
11. Subjects with symptomatic brain metastases, or with any symptoms suggestive of brain metastases or intracranial hypertension;
12. With uncontrolled serosal effusion;
13. Patients with serious cardiovascular diseases;
14. Concurrent uncontrolled hypertension before randomization;
15. Patients with active hepatitis B, active hepatitis C, acquired immunodeficiency syndrome (AIDS) or HIV test positive, and active syphilis test positive;
16. Concomitant diseases where dexamethasone is contraindicated;
17. The presence of severe or inadequately controlled diseases;
18. Known contraindications to NK-1 receptor antagonists, 5-HT3 receptor antagonists, or dexamethasone;
19. Participation in another clinical trial within 30 days prior to randomization (based on the use of study medication);
20. The presence of severe emotional or psychiatric disorders, as assessed by the investigator as unsuitable for participation in this study;
21. Subjects who, in the opinion of the investigator, have other conditions that make them inappropriate for participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 706 (Actual)
Dates: Start 2024-09-03 (Actual); Primary Completion 2025-07-28 (Actual); Study Completion 2025-10-03 (Actual)

PRIMARY OUTCOMES:
Complete response rate in the delayed phase | 24-120 hours after initiation of moderate emetic risk anticancer agents
  To compare the rate of subjects achieving complete response (defined as no emetic episode and no need for rescue medication) in the delayed phase after initiation of moderate emetic risk anticancer agents.

SECONDARY OUTCOMES:
Complete response rate in the overall phase. | 0 - 120 hours after initiation of moderate emetic risk anticancer agents
  To compare the rate of subjects achieving complete response (defined as no emetic episode and no need for rescue medication) in the overall phase after initiation of moderate emetic risk anticancer agents.
Complete response rate in the acute phase. | 0-24 hours after initiation of moderate emetic risk anticancer agents
  To compare the rate of subjects achieving complete response (defined as no emetic episode and no need for rescue medication) in the acute phase after initiation of moderate emetic risk anticancer agents.
Proportion of subjects with no significant nausea (maximum nausea on a visual analogue scale<25 mm) | the acute phase (0-24 hours), the delayed phase(24 - 120 hours), and the overall phase (0-120 hours) after initiation of moderate emetic risk anticancer agents, respectively
  To compare the proportion of subjects achieving no significant nausea (defined as maximum nausea on a visual analogue scale<25 mm) in the acute phase (0-24 hours), the delayed phase(24 - 120 hours), and the overall phase (0-120 hours) after initiation of moderate emetic risk anticancer agents, respectively
Proportion of subjects with no nausea (maximum nausea on a visual analogue scale<5 mm) | the acute phase (0-24 hours), the delayed phase(24 - 120 hours), and the overall phase (0-120 hours) after initiation of moderate emetic risk anticancer agents, respectively
  To compare the proportion of subjects achieving no nausea (defined as maximum nausea on a visual analogue scale<5 mm) in the acute phase (0-24 hours), the delayed phase(24 - 120 hours), and the overall phase (0-120 hours) after initiation of moderate emetic risk anticancer agents, respectively
Proportion of subjects with no emetic | the acute phase (0-24 hours), the delayed phase(24 - 120 hours), and the overall phase (0-120 hours) after initiation of moderate emetic risk anticancer agents, respectively
  To compare the proportion of subjects with no emetic event in the acute phase (0-24 hours), the delayed phase(24 - 120 hours), and the overall phase (0-120 hours) after initiation of moderate emetic risk anticancer agents, respectively
Proportion of subjects with no rescue medication | the acute phase (0-24 hours), the delayed phase(24 - 120 hours), and the overall phase (0-120 hours) after initiation of moderate emetic risk anticancer agents, respectively
  To compare the proportion of subjects with no rescue medication in the acute phase (0-24 hours), the delayed phase(24 - 120 hours), and the overall phase (0-120 hours) after initiation of moderate emetic risk anticancer agents, respectively
Proportion of subjects with complete protection | the acute phase (0-24 hours), the delayed phase(24 - 120 hours), and the overall phase (0-120 hours) after initiation of moderate emetic risk anticancer agents, respectively
  To compare the proportion of subjects achieving complete protection (defined as no emetic episode, no significant nausea and no need for rescue medication) in the acute phase (0-24 hours), the delayed phase(24 - 120 hours), and the overall phase (0-120 hours) after initiation of moderate emetic risk anticancer agents, respectively
Proportion of subjects with total control | the acute phase (0-24 hours), the delayed phase(24 - 120 hours), and the overall phase (0-120 hours) after initiation of moderate emetic risk anticancer agents, respectively
  To compare the proportion of subjects achieving total control (defined as no emetic episode, no nausea and no need for rescue medication) in the acute phase (0-24 hours), the delayed phase (24 - 120 hours), and the overall phase (0-120 hours) after initiation of moderate emetic risk anticancer agents, respectively
Time to treatment failure | 0-120 hours after initiation of moderate emetic risk anticancer agents
  Time to the first occurrence of emetic event or the first rescue medication
The score using the functional living index-emesis (FLIE) questionnaire | 0-120 hours after initiation of moderate emetic risk anticancer agents
  Changes in the score of FLIE before and after treatment
Adverse events | Approximately 4 weeks
  To analyse the rates of adverse events as assessed by CTCAE v5.0

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center Yuexiu Campus, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided